CLINICAL TRIAL: NCT06332833
Title: Availability of Venous Conduits in Patients With Varicose Veins for Arterial Bypass Surgery
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 235
Record Dates: First submitted 2024-03-15; First posted 2024-03-27 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2023-12

CONDITIONS: Varicose Veins; Peripheral Arterial Disease
Keywords: varicose veins; Peripheral Arterial Disease; phlebectomy
MeSH Terms: conditions — Varicose Veins; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with PAD having superficial femoral artery (SFA) occlusion were consecutively enrolled. Demographic data and medical history were taken. Physical examination and duplex ultrasound were performed.

DETAILED DESCRIPTION:
Patients with PAD having superficial femoral artery (SFA) occlusion were consecutively enrolled. Demographic data and medical history were taken. Physical examination and duplex ultrasound were performed. The investigators registered presence of varicose veins, type of previous invasive procedure and availability of saphenous trunks as possible grafts

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 Years

Exclusion Criteria:

* Those unwilling to sign an informed consent were also included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PAD having superficial femoral artery (SFA) occlusion.
Sampling Method: Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
availability of saphenous trunks as possible grafts | at the moment of inclusion
  availability of saphenous trunks as possible grafts (Yes|No)

SECONDARY OUTCOMES:
presence of varicose veins | at the moment of inclusion
  presence of varicose veins (Yes|No)
type of previous invasive procedure | at the moment of inclusion
  Phlebectomy\ radiofrequency ablation\ endovenous laser ablation (Yes|No)

CONTACTS AND LOCATIONS:
Locations (1):
- Veronika Golovina, Moscow, Pirogov Russian National Research Medical University, Russia